CLINICAL TRIAL: NCT06697652
Title: Early Readmission After Adrenalectomy for PHEO.
Brief Title: Readmission After Adrenalectomy
Status: Completed | Type: Observational
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Tamer.A.A.M.Habeeb, prof, Zagazig University
Other Study IDs: early readmission after pheo s
Record Dates: First submitted 2024-11-18; First posted 2024-11-20 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Adrenalectomy
Keywords: adrenalectomy; hospital; risk factors
MeSH Terms: interventions — Adrenalectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- hospital readmission: hospital readmission for complications
  Interventions: Procedure: adrenalectomy

INTERVENTIONS:
Procedure: adrenalectomy — adrenalectomy

SUMMARY:
to evaluate early hospital enterance after pheo surg.

ELIGIBILITY:
Inclusion Criteria:

* patients with pheo

Exclusion Criteria:

* non reactive
* missed data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with pheo
Sampling Method: Non-Probability Sample
Enrollment: 346 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2024-09-01 (Actual)

PRIMARY OUTCOMES:
readmission rate | 30 days
  number of hospital readmission

IPD SHARING:
Plan to Share IPD: Undecided